CLINICAL TRIAL: NCT04392973
Title: A Trial of Favipiravir and Hydroxychloroquine Combination in Adults Hospitalized With Moderate and Severe Covid-19
Brief Title: FAvipiravir and HydroxyChloroquine Combination Therapy
Acronym: FACCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah International Medical Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC20/174
Record Dates: First submitted 2020-05-10; First posted 2020-05-19 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: COVID19
Keywords: SARS-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — favipiravir; Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: Randomized, open-label, parallel groups were participants are assigned to either an intervention arm or standard of care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Combination therapy Favipiravir (10 days) + Hydroxychloroquine(5 days)
  Interventions: Combination Product: Favipiravir and Hydroxychloroquine
- Control (No Intervention): Standard of Care Treatment for COVID-19 Infection

INTERVENTIONS:
Combination Product: Favipiravir and Hydroxychloroquine — Route of Administration: Oral (or through Nasogastric tube)
  Dose:
  Favipiravir: Administer 1800 mg (9 tablets) by mouth twice daily for one day, followed by 800mg (4 tablets) twice daily (total days of therapy is 10 days or till hospital discharge)
  Hydroxychloroquine (400mg) twice daily on day 1; for days 2-5 (200mg) twice daily.
  Other Names: Avigan
  Arms: Intervention

SUMMARY:
This study is a randomized, open-label, parallel groups multi-centered trial were participants are assigned to either an intervention arm ( a combination of Favipiravir and Hydroxychloroquin) or standard of care.

DETAILED DESCRIPTION:
In this trial, the investigators want to evaluate the efficacy of the combination of Favipiravir and Hydroxychloroquine as potential therapy for moderate and severe cases with COVID -19. Favipiravir which is a new type of RNA-dependent RNA polymerase (RdRp) inhibitor has activity against influenza virus, and Hydroxychloroquine, an analogue of chloroquine, has a clinical safety profile better than that of chloroquine and allows higher daily dose, Chloroquine is a widely used antimalarial that was found to be a potential broad-spectrum antiviral.

There is an urgent need to explore therapeutic options for SARS-CoV-2 in order to face the pandemic. The selected combination was based on limited evidence clinically and in vitro on the efficacy of the Favipiravir and Hydroxychloroquine in SARS-CoV-2. The two medications were listed in many guidelines as treatment options and ongoing trials assessing their efficacy and safety. Thus, the investigators want to prove the effectiveness of the combination as therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Should be at least 18 years of age
2. Male or nonpregnant female,
3. Diagnosed with COVID-19 by PCR confirmed SARS-coV-2 viral infection.
4. Able to sign the consent form and agree to clinical samples collection (or their legal surrogates if subjects are or become unable to make informed decisions).
5. Moderate or Severe COVID-19, defined as oxygen saturation (Sao2) of 94% or less while they were breathing ambient air or significant clinical symptoms with Chest X ray changes that require hospital admission.
6. patients had to be enrolled within 10 days of disease onset

Exclusion Criteria:

1. Patients who are pregnant or breastfeeding.
2. Will be transferred to a non-study site hospital or expected to be discharged within 72 hours.
3. Known sensitivity/allergy to hydroxychloroquine or Favipiravir
4. Current use of hydroxychloroquine for another indication
5. Prior diagnosis of retinopathy
6. Prior diagnosis of glucose-6-phosphate dehydrogenase (G6PD) deficiency
7. Major comorbidities increasing the risk of study drug including: i. Hematologic malignancy, ii. Advanced (stage 4-5) chronic kidney disease or dialysis therapy, iii. Known history of ventricular arrhythmias, iv. Current use of drugs that prolong the QT interval, Severe liver damage (Child-Pugh score ≥ C, AST> 5 times the upper limit), HIV.
8. The investigator believes that participating in the trial is not in the best interests of the patient, or the investigator considers unsuitable for enrollment (such as unpredictable risks or subject compliance issues).
9. Clinical prognostic non-survival, palliative care, or in deep coma and no have response to supportive treatment within three hours of admission.
10. Patient with irregular rhythm
11. Patient with a history of heart attack (myocardial infarction)
12. Patient with a family history of sudden death from heart attack before the age of 50
13. Take other drugs that can cause prolonged QT interval
14. Patient who is receiving immunosuppressive therapy (cyclosporin) which cannot be switched to another agent or adjusted while using the investigational drug
15. Gout/history of Gout or hyperuricemia (above the ULN), hereditary xanthinuria or xanthine calculi of the urinary tract.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2020-05-21 (Actual); Primary Completion 2021-01-26 (Actual); Study Completion 2021-04-26 (Actual)

PRIMARY OUTCOMES:
Clinical Improvement | 28 days
  The primary endpoint is the time to clinical improvement, defined as the time from the randomization to an improvement of two points (from the status at randomization) on a seven-category ordinal scale or live discharge from the hospital, whichever came first.

SECONDARY OUTCOMES:
Viral shedding | 28 days
  PCR test negative conversion days from positive to negative.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Alaskar, Study Director — KAIMRC
Locations (8):
- Saudi Arabia (8):
  - King Abdulaziz Hospital - Al Ahsa, Hasa, Eastern Province
  - AlMadina General Hospital, Al Madīnah
  - Al-Qatif Central Hospital, Al Qaţīf
  - Imam Abdulrahman Al Faisal Hospital - Dammam, Dammam
  - King Abdulaziz Medical City, Jeddah
  - King Abdulaziz Hospital - Makkah, Mecca
  - King Abdulaziz Medical City, National Guard Health Affairs, Riyadh
  - Imam Abdulrahman Alfaisal Hospital, Riyadh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bosaeed M, Mahmoud E, Alharbi A, Altayib H, Albayat H, Alharbi F, Ghalilah K, Al Arfaj A, AlJishi J, Alarfaj A, Alqahtani H, Almutairi BM, Almaghaslah M, Alyahya NM, Bawazir A, AlEisa S, Alsaedy A, Bouchama A, Alharbi M, AlShamrani M, Al Johani S, Aljeraisy M, Alzahrani M, Althaqafi AO, Almarhabi H, Alotaibi A, Alqahtani N, Arabi YM, Aldibasi OS, Alaskar A. Favipiravir and Hydroxychloroquine Combination Therapy in Patients with Moderate to Severe COVID-19 (FACCT Trial): An Open-Label, Multicenter, Randomized, Controlled Trial. Infect Dis Ther. 2021 Dec;10(4):2291-2307. doi: 10.1007/s40121-021-00496-6. Epub 2021 Jul 28. PMID 34319552
- [Derived] Bosaeed M, Mahmoud E, Hussein M, Alharbi A, Alsaedy A, Alothman A, Aljeraisy M, Alqahtani H, Nashabat M, Almutairi B, Almaghaslah M, Aldibasi O, AlJohani S, Bouchama A, Arabi Y, Alaskar A. A Trial of Favipiravir and Hydroxychloroquine combination in Adults Hospitalized with moderate and severe Covid-19: A structured summary of a study protocol for a randomised controlled trial. Trials. 2020 Oct 31;21(1):904. doi: 10.1186/s13063-020-04825-x. PMID 33129363